CLINICAL TRIAL: NCT02298101
Title: Comparison of Lung Deposition With the Aeroneb Solo Adapter and a Standard Jet Nebulizer by SPECT-CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AeroSpect-01
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Aerosol delivery; Lung deposition; SPECT; subjects
MeSH Terms: interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Aeroneb Solo Adapter (Active Comparator): Subjects inhaled radiolabelled aerosol via the Aeroneb Solo Adapter
  Interventions: Drug: Technetium-99m - Diethylenetriaminepentaacetic acid; Device: Aeroneb Solo Adapter; Other: Planar scintigraphy; Other: Single photon emission computed tomography; Other: Spirometry
- Standard Jet Nebulizer (Active Comparator): Subjects inhaled radiolabelled aerosol via a standard jet nebulizer, the Opti-Mist Plus Nebulizer
  Interventions: Drug: Technetium-99m - Diethylenetriaminepentaacetic acid; Device: Opti-Mist Plus Nebulizer; Other: Planar scintigraphy; Other: Single photon emission computed tomography; Other: Spirometry

INTERVENTIONS:
Drug: Technetium-99m - Diethylenetriaminepentaacetic acid — Solution placed on the nebulizer reservoir
Device: Aeroneb Solo Adapter — Nebulizer
  Arms: Aeroneb Solo Adapter
Device: Opti-Mist Plus Nebulizer — Standard jet nebulizer
  Arms: Standard Jet Nebulizer
Other: Planar scintigraphy — Imaging technique to investigate whole lung deposition
Other: Single photon emission computed tomography — Imaging technique to investigate regional pulmonary deposition
Other: Spirometry — FEV1, FVC assessment

SUMMARY:
Aeroneb Solo Adapter is a vibrating-mesh nebulizer Aeroneb Solo combined to a spacer specifically designed for spontaneously breathing patients. This device has not been investigated in vivo yet.

It's known that using a spacer during nebulization improves aerosol delivery. We hypothetized that lung deposition could be highly increased with the Aeroneb Solo Adapter in comparison to a standard jet nebulizer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy respiratory function

Exclusion Criteria:

* Pulmonary disease

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary deposition | immediately after nebulization by imaging assessment, an expected average of 15 minutes
  Planar scintigraphy and single photon emission computed tomography as imaging techiques

SECONDARY OUTCOMES:
Three-dimensional penetration index | immediately after the nebulization by imaging assessment, expected average of 30 minutes
  Single photon emission computed tomography as imaging technique

OTHER OUTCOMES:
Spirometry | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Dugernier J, Hesse M, Vanbever R, Depoortere V, Roeseler J, Michotte JB, Laterre PF, Jamar F, Reychler G. SPECT-CT Comparison of Lung Deposition using a System combining a Vibrating-mesh Nebulizer with a Valved Holding Chamber and a Conventional Jet Nebulizer: a Randomized Cross-over Study. Pharm Res. 2017 Feb;34(2):290-300. doi: 10.1007/s11095-016-2061-7. Epub 2016 Nov 7. PMID 27822851